CLINICAL TRIAL: NCT00980915
Title: Identifying Patients at Risk of Developing Acute Lung Injury at the Time of Hospital Admission:Toward the Prevention of Acute Lung Injury (ALI)
Brief Title: Timing and Intensity of the Exposures and Attributable Burden of Acute Lung Injury
Acronym: LIPS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, Ognjen Gajic, M.D., Mayo Clinic
Other Study IDs: 08-003560; LIPSSTUDY
Record Dates: First submitted 2009-04-30; First posted 2009-09-21 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: Acute Lung Injury; Acute Respiratory Distress Syndrome; Respiratory Distress; pneumonia; sepsis; aspiration; pancreatitis
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome; Dyspnea; Pneumonia; Sepsis; Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will collect time sensitive peripheral blood samples for collaborative genome-wide association, gene expression, cytokines and proteonomic studies. Blood samples of the enrolled patients will be collected as baseline, after 24, 48 hours and at the time of development of ARDS.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- At risk for Acute Lung Injury: Controls-High risk patients at risk of Acute Lung Injury(ALI) but do not develop ALI
  Cases-High risk patients that do develop Acute Lung Injury

SUMMARY:
The purpose of the study is to identify the patients at high risk of developing Acute Lung Injury (ALI) at the time of hospital admission, and before intensive care unit admission.

Aim 1- To validate the prediction model (Lung Injury Prediction Score) in a population based sample of hospitalized patients.

Aim 2- To determine the significance of health-care related ALI risk modifiers in a population based sample.

Aim 3- To compare the short and long term outcomes between patients at high risk who do, and do not develop ALI.

DETAILED DESCRIPTION:
Acute lung injury (ALI) is an example of a critical care syndrome with limited treatment options once the condition is fully established.Not surprisingly, many treatments targeting the mechanisms identified in preclinical studies have failed to improve patient outcomes.The most likely reason could be due to inadequate and delayed recognition of patients at risk and the subsequent development of the full blown syndrome.ALI/ARDS usually develops during the first hours of ICU admission, and often is the very reason for ICU admission.

Clinical prediction models have been extensively used in the clinical practice to identify patients at high risks who may benefit from specific interventions. However, no such tool exists to predict the development of ALI in patients at risk. We have recently developed an ALI prediction model (Lung Injury Prediction Score:LIPS)which incorporates demographic, environmental and clinical characteristics at the time of, and before, hospital admission. If validated, this model will serve to find the population of patients at high risk of ALI in whom future prevention trials will be conducted. By determining not only patients at high risk but also the attributable burden of ALI/ARDS in contemporary cohorts of patients at risk, our findings will facilitate the prioritization of preventive strategies and future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* All Olmsted County residents more than 18 years of age who were admitted to the two Mayo Clinic Rochester hospitals

Exclusion Criteria:

* Denied the use of medical records for research
* Acute lung injury or pulmonary edema already present at the time of hospital admission
* Admitted for comfort or hospice care only
* Children
* Hospital readmission
* Patients admitted for cardiac telemetry, coronary care unit, low risk elective surgeries, labor and delivery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Olmsted County residents more than 18 years of age who were admitted to the two Mayo Clinic Rochester hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 6600 (Estimated)
Dates: Start 2008-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Development of ALI | During the hospital stay (before discharge and maximum of 30 days)

SECONDARY OUTCOMES:
Quality adjusted survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ognjen Gajic, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials